CLINICAL TRIAL: NCT01275612
Title: Ex-Vivo Expanded Mesenchymal Stem Cells To Repair The Kidney And Improve Function In Cisplatin-Induced Acute Renal Failure In Patients With Solid Organ Cancers
Brief Title: Mesenchymal Stem Cells In Cisplatin-Induced Acute Renal Failure In Patients With Solid Organ Cancers
Acronym: CIS/MSC08
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Patients evaluated so far could not be enrolled because they did not meet the primary criterion of acute renal failure provided by the study protocol
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIS/MSC 08; 2008-007485-35 (EudraCT Number)
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Solid Tumors; Acute Kidney Injury
Keywords: Mesenchymal Stromal Cells; Solid tumors; Cisplatin therapy; Acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cell therapy (Experimental)
  Interventions: Biological: Mesenchymal stromal cell infusion

INTERVENTIONS:
Biological: Mesenchymal stromal cell infusion — The first 3 patients will receive a single i.v infusion of donor ex-vivo expanded MSC (1 x 106 MSC/kg). If the efficacy outcome of cell treatment is negligible or partial and the procedure is safe, a second group of additional 3 patients will be enrolled. They will be given MSC i.v infusion at higher dose (2 x 106 MSC/kg).Should the therapeutic efficacy of this treatment again negligible or marginal, but still safe, a third group of 3 patients will be enrolled in the study. The dose of cells to be infused will be up-titrated to 5 x 106 MSC/kg.

SUMMARY:
This is a pilot, explorative, study to test the feasibility and safety of systemic infusion of donor ex-vivo expanded Mesenchymal Stem Cells to repair the kidney and improve function in patients with solid organ cancers who develop acute renal failure after chemotherapy with cisplatin.

DETAILED DESCRIPTION:
Since its introduction into clinical trials, cisplatin (cis-diammine-dichloro-platinum) has had a major impact in cancer medicine, changing the course of therapeutic management of several tumors, such as those of ovary, testes, and the head and neck. Unfortunately, in addition to causing bone marrow suppression, ototoxicity, and anaphylaxis, dose-dependent and cumulative nephrotoxicity is the major toxicity of this compound, sometimes requiring a reduction in dose or discontinuation of treatment. Approximately 25-35% of patients develop evidence of nephrotoxicity following an initial dose (50-100 mg/m2) of cisplatin, due to its preferential accumulation within the proximal tubular cells in the outer medulla of the kidney. Tubular cell events activated by cisplatin toxicity translate into the fact that cisplatin predictably lowers glomerular filtration rate (GFR) in a clear dose-dependent manner even after a single drug exposure. Early proteinuria is mild, as it is glycosuria. Overall these findings indicate that there is a pressing need for way to protect the kidney while administering effective chemotherapeutic agents such as cisplatin.

Present strategies for the treatment of acute renal failure have focused on targeting individual mechanisms thought to contribute to ischemic or toxic insults to the kidney.An alternative possibility is to adopt a novel strategy that would allow regeneration of the injured renal tissue. Renal recovery following acute tubular injury, like that induced by cisplatin treatment, is often a slow process requiring many days to weeks to occur. Attempts to accelerate recovery have focused on the administration of growth factors, hepatocyte growth factor, or insulin-like growth factor-1. While growth factor therapy has been successful in experimental models, no beneficial effects have been observed in limited clinical trials. The ability of extrarenal cells to participate in the regenerative response following post-transplant acute renal failure may hold true for acute renal failure that develops in native kidneys after cisplatin therapy. The rationale for this approach rests on the recent demonstration in mice and in athymic nude rats that stem cells from bone marrow can be used to grow new muscle or blood vessels in heart tissue that has been damaged after myocardial infarction. Similarly, consistent evidence of the beneficial effect of bone-marrow derived cell therapy has been recently reported in humans with ischemic heart disease. This approach has been also successfully extended to repair ischemically and cisplatin injured renal tubules in mice. The observation raises the possibility that adult-derived bone marrow cells could be administered to enhance the recovery from renal injury. Although no human data so far are available, we expect that ex-vivo expanded donor bone-marrow derived mesenchymal stromal cells (MSC) infusion would allow to accelerate tubular regeneration and thus renal function recovery in patients with cisplatin-induced acute renal failure, a disease that, like ischemically-induced acute renal injury, so far has no cure.

Up to now there is no clinical study of repair tissue injury in patients with acute renal failure due to ischemic or toxic insults. Nevertheless, there are clinical data on the effectiveness of MSC infusion in other diseases/conditions like as inborn errors of metabolism,osteogenesis imperfecta,allogeneic HSC transplantation, treatment of acute GVHD, acute myocardial infarction.

The aim of this pilot, explorative, study is to test the feasibility and safety of systemic infusion of donor ex-vivo expanded MSC to repair the kidney and improve function in patients with solid organ cancers who develop acute renal failure after chemotherapy with cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Requiring cisplatin therapy (>80mg/m2) against advanced head and neck carcinoma, non-small cell lung cancer stage IIIB/IV, bladder transitional cell carcinoma locally advanced or metastatic, which are not amenable to surgical resection or ablation with curative intent
* An Eastern Cooperative Oncology Group performance status (ECOG PS) <2
* Normal renal, hepatic and bone marrow function
* Physician's assessment of life expectancy: 4-10 months
* Aged > 18 years
* Evidence of acute renal injury as assessed by percent increase of NGAL concentration in spot urine > 3500% over baseline values at day 2 post-cisplatin infusion
* Written informed consent

Exclusion Criteria:

* Specific contraindication to MSC infusion
* Serious concomitant diseases not adequately responding to specific therapy
* Symptomatic brain metastases
* Pregnancy
* Previous cisplatin infusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Serum creatinine concentration. | 15 days post-cisplatin infusion
  To evaluate the rate of renal function loss up to 15 days post-cisplatin infusion.

SECONDARY OUTCOMES:
Neutrophil gelatinase-associated lipocalin (NGAL) | At days 0,2,5,7,12,15,18 and 30.
N-acetyl-p- D glucosaminidase enzyme (NAG) | At days 0,2,5,7,12,15,18 and 30.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Chair — Department of Immunology and Clinical Transplantation/Mario Negri Institute for Pharmacological Research and Ospedali Riuniti of Bergamo; Norberto Perico, MD, Principal Investigator — Mario Negri Institute for Pharmacological Research; Martino Introna, MD, Principal Investigator — Cell and Gene Therapy Laboratory "G.Lanzani" Bergamo; Alessandro Rambaldi, MD, Principal Investigator — Unit of Hematology - Ospedali Riuniti of Bergamo; Carlo Tondini, MD, Principal Investigator — Unit of Oncology - Ospedali Riuniti of Bergamo
Locations (1):
- Unit of Oncology - Ospedali Riuniti of Bergamo, Bergamo, BG, Italy